CLINICAL TRIAL: NCT07359690
Title: Multimodal Analysis of Endomyocardial Biopsies
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Lars Michel, Head of Cardiomyopathies and Heart Failure, University Hospital, Essen
Other Study IDs: WHGZ-EMB
Record Dates: First submitted 2025-12-16; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation; Dilated Cardiomyopathy (DCM); Hypertrophic Cardiomyopathy (HCM); Myocarditis, Pericarditis; Amyloidosis Cardiac; Cardiomyopathies; Sarcoidosis of the Heart
Keywords: Endomyocardial biopsy; Multimodal analysis
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Myocarditis; Pericarditis; Amyloid Neuropathies, Familial; Cardiomyopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Endomyocardial biopsy samples containing DNA for further multi-omics assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing endomyocardial biopsy following clinical indication: All patients with a clinical indication for EMB without regard to certain disease types. Typically these patients are after heart transplantation, amyloidosi or with a cardiomyopathy, including dilated-, hypertrophic- or inflammatory cardiomyopathy.

SUMMARY:
The goal of this observational study is to pursue a multimodal approach to identify the molecular signatures and immune signalling molecules of various myocardial diseases and thereby contribute to improving diagnosis and therapy.

The main aim is:

-Identification of molecular profiles (e.g., proteome, lipidome, metabolome) and immune signalling profiles that are specifically associated with different myocardial diseases and the post-heart transplantation course.

Participants already receiving an endomyocardial biopsy as part of their regular medical care will be enrolled. An additional biopsy sample will be taken for the above mentioned research.

DETAILED DESCRIPTION:
The proposed study aims to pursue a multimodal approach to identify the molecular signatures and immune signalling profiles of various myocardial diseases and thereby contribute to improving diagnosis and therapy. In the context of a clinically indicated endomyocardial biopsy (EMB), an additional EMB will be performed. This sample will be further analyzed using, among other methods, multi-omics, immune signalling analysis and nuclear cardiology analyses. These analyses are intended to enable the identification of genetic mutations, inflammatory gene expression patterns, immune signalling and protein alterations in myocardial diseases such as cardiomyopathies, myocarditis, and cardiac amyloidosis. Furthermore, the results will be correlated with established clinical parameters and biomarkers in order to identify novel diagnostic markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years with a clinical indication for endomyocardial biopsy.
* Patients capable of providing informed consent who have signed the consent form for participation in the study.

Exclusion Criteria:

* Patients without a clinical indication for endomyocardial biopsy (EMB).
* Pregnant individuals.
* Patients incapable of providing informed consent.
* Women of childbearing potential who are not using adequate contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients receiving an endomyocardial biopsy after routine clinical indication will be enrolled. The identification of molecular profiles from the obtained endomyocardial biopsies (EMBs) represents an exploratory research approach that does not allow for an exact sample size calculation. Considering the heterogeneity of the collected EMBs, and particularly the fact that EMBs are often performed for the differential diagnosis of various rare myocardial diseases, an adequately large study population is necessary to capture rare phenotypes. The planned cohort will include 40 patients each from the main groups: unclear cardiomyopathy, suspected (ICI-)myocarditis, suspected cardiac storage disease, and post-heart transplantation surveillance. Thus, a total of 160 EMBs are targeted for multi-omics analysis.The secondary endpoint of the study allows for a sample size estimation of 56 EMBs for the subgroup of cardiac amyloidosis (calculation according to the full proposal).
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Spatial molecular profiles and immune signalling in all included patients | Baseline, up to 1 year
  Identification of spatial molecular profiles (e.g., proteomic, lipidomic, and metabolomic signatures) and immune signalling pathways specifically associated with various myocardial diseases and post-heart transplantation outcomes.

SECONDARY OUTCOMES:
Tracer-Uptakes in cardiac amyloidosis. | Baseline, up to 1 year.
  Ex vivo analysis of tracer uptake in human endomyocardial biopsy samples from patients with cardiac amyloidosis.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Michel, PD Dr. med., Principal Investigator — Department of Cardiology and Vascular Medicine, West German Heart and Vascular Center Essen, University Hospital Essen, Germany
Locations (1):
- Department of Cardiology and Vascular Medicine, West German Heart and Vascular Center Essen, University Hospital Essen, Germany, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided